CLINICAL TRIAL: NCT07084259
Title: HArnessing Near-infrared Spectroscopy Intravascular Ultrasound Imaging for Yielding Advanced Guidance - PCSK9i for Improving Cardiovascular Outcome in High-Risk Patients
Brief Title: Single Dose PCSK9 Inhibitor to Improve Cardiovascular Outcomes After PCI: A Pilot Study
Acronym: HANYANG-PICK
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Hanyang University Seoul Hospital (Other)
Collaborators: DOTTER Inc. (Unknown)
Responsible Party: Principal Investigator, Woohyeun Kim, Associate Professor, Division of Cardiology, Department of Internal Medicine, Hanyang University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HYUH 2025-02-018-004
Record Dates: First submitted 2025-07-16; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Coronary Artery Disease
Keywords: PCSK9 Inhibitor; Near-Infrared Spectroscopy (NIRS); Intravascular Ultrasound (IVUS); Vulnerable Plaque; Evolocumab
MeSH Terms: conditions — Coronary Artery Disease | interventions — evolocumab

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned in a parallel manner to receive either a PCSK9 inhibitor (Evolocumab) in addition to standard therapy or standard therapy alone. The study aims to compare the long-term cardiovascular outcomes between the two groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PCSK9 Inhibitor Group (Experimental): Patients with elevated post-PCI LCBI receiving a single subcutaneous dose of a PCSK9 inhibitor (evolocumab 140 mg) after percutaneous coronary intervention.
  Interventions: Drug: PCSK9 inhibitor
- Standard of Care Group (Active Comparator): Patients receiving standard post-PCI treatment without PCSK9 inhibitor therapy. Lipid-lowering therapy is managed according to current clinical guidelines.
  Interventions: Drug: Standard Lipid-Lowering Therapy

INTERVENTIONS:
Drug: PCSK9 inhibitor — Single dose of subcutaneous administration of PCSK9 inhibitors (evolocumab) after PCI in patients with coronary artery disease and elevated post-PCI lipid core burden (maxLCBI4mm ≥ 200).
  Other Names: Evolocumab (Repatha)
  Arms: PCSK9 Inhibitor Group
Drug: Standard Lipid-Lowering Therapy — Lipid-lowering therapy with high-intensity or maximally tolerated statins with or without ezetimibe, as per current clinical guidelines, excluding the use of PCSK9 inhibitors.
  Other Names: Statins ± Ezetimibe
  Arms: Standard of Care Group

SUMMARY:
This pilot study aims to evaluate whether a single dose of PCSK9 inhibitor administered after percutaneous coronary intervention (PCI) can improve long-term cardiovascular outcomes in patients with high post-PCI lipid core burden, as assessed by NIRS-IVUS. The study will assess major adverse cardiovascular events (MACE) over a 12-month follow-up period.

DETAILED DESCRIPTION:
Coronary artery disease (CAD) remains a leading cause of death worldwide, and while PCI has improved clinical outcomes, residual cardiovascular risk persists, especially in patients with lipid-rich plaques. Near-infrared spectroscopy combined with intravascular ultrasound (NIRS-IVUS) allows for the detection of lipid core burden, and high post-PCI LCBI values have been associated with worse prognosis.

This single-center, prospective, randomized pilot study (HANYANG-PICK) investigates the impact of a single dose of PCSK9 inhibitor administered immediately after PCI in patients with high post-PCI LCBI. The intervention group will receive the PCSK9 inhibitor, and the control group will undergo standard therapy. The primary endpoint is the incidence of major adverse cardiovascular events (MACE) at 12 months. The study is designed to inform the feasibility of a larger trial and to explore the potential of PCSK9 inhibitors for early plaque stabilization post-PCI.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 19 years or older
* Patients diagnosed with coronary artery disease, including silent ischemia, stable angina, or acute coronary syndrome (unstable angina, NSTEMI, or STEMI)
* Underwent percutaneous coronary intervention (PCI) with NIRS-IVUS imaging
* Presence of target vessel post-PCI maxLCBI4mm ≥ 200
* Able and willing to provide written informed consent

Exclusion Criteria:

* Cardiogenic shock or hemodynamic instability within 24 hours prior to enrollment
* Expected life expectancy <1 year
* Participation in another investigational study that may interfere with the results
* Known contraindications to PCSK9 inhibitors or standard-of-care lipid-lowering therapy

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 352 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2030-06 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
Patient-oriented Composite Outcome (MACE) | 12 months
  Composite of all-cause mortality, any myocardial infarction, any stroke, or any clinically driven revascularization.

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) will be made available upon reasonable request to qualified researchers. The data will be made available following publication of the primary results upon request and will be available for 5 years.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: IPD and supporting information will be available beginning 12 months after publication of the primary results and will remain available for up to 5 years, contingent upon approval by the HANYANG-PICK Steering Committee.
Access Criteria: Access to the de-identified individual participant data (IPD) and supporting documents will be granted to qualified researchers who submit a methodologically sound proposal, as determined by the HANYANG-PICK Steering Committee. The proposed research must be for non-commercial, academic purposes. Requestors will be required to sign a data use agreement and obtain appropriate ethical approvals before accessing the data.